CLINICAL TRIAL: NCT00890708
Title: Influence of Therapeutic Drug Monitoring of Voriconazole on Incidence of Drug Adverse Reaction
Brief Title: Therapeutic Drug Monitoring of Voriconazole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wan Beom Park, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-0808-057-254
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Mycoses
MeSH Terms: conditions — Mycoses | interventions — Voriconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- non-TDM of voriconazole (No Intervention): conventional dose
- TDM of voriconazole (Experimental)
  Interventions: Drug: Voriconazole (therapeutic drug monitoring)

INTERVENTIONS:
Drug: Voriconazole (therapeutic drug monitoring) — dosage adjustment according to trough level of voriconazole in plasma
  Other Names: plasma drug level
  Arms: TDM of voriconazole

SUMMARY:
The purpose of this study is to determine whether therapeutic drug monitoring of voriconazole is useful in the treatment of invasive fungal infection.

DETAILED DESCRIPTION:
Voriconazole is an anti-fungal agent, which is used in the treatment of invasive fungal infection, especially aspergillosis. The serious side effects of voriconazole include liver function abnormality, encephalopathy, etc. Recently, the several studies showed that the blood level of voriconazole is variable and it is associated with drug side effect and treatment outcome. However, there is no randomized controlled study which proves that therapeutic drug monitoring of voriconazole can improve the clinical outcome in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients who were 16 years of age or older
* receiving voriconazole in order to treat invasive fungal infections or for empirical use

Exclusion Criteria:

* who experienced the serious side effect of voriconazole
* were hypersensitive to azoles
* had an aminotransferase, bilirubin, or alkaline phosphatase level higher than five times the upper limit of normal

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
side effects | during 3 months

SECONDARY OUTCOMES:
treatment response to voriconazole | at 3 months
drug discontinuation of adverse events | within 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Wan Beom Park, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park WB, Kim NH, Kim KH, Lee SH, Nam WS, Yoon SH, Song KH, Choe PG, Kim NJ, Jang IJ, Oh MD, Yu KS. The effect of therapeutic drug monitoring on safety and efficacy of voriconazole in invasive fungal infections: a randomized controlled trial. Clin Infect Dis. 2012 Oct;55(8):1080-7. doi: 10.1093/cid/cis599. Epub 2012 Jul 3. PMID 22761409